CLINICAL TRIAL: NCT04507100
Title: Comprehensive Analysis of the Program:Salud Escolar
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial twithdrawn due to the COVID-19 pandemic
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: UNICEF (Other); Ministry of Education, Mexico (Other Government); Ministry of Health, Mexico (Unknown)
Responsible Party: Principal Investigator, Alejandra Jáuregui de la Mota, Chair of the Department of Physical Activity and Healthy Lifestyles, Instituto Nacional de Salud Publica, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P86-19
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Obesity
Keywords: physical activity; healthy eating; hydration; school intervention; health policy
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Masking Description: Masking is not possible because the Ministry of Education specifically announces the implementation of Salud Escolar in each school.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle and environment intervention (Experimental): Schools will receive the components of Salud Escolar
  Interventions: Behavioral: World Health Organization Health Promoting Schools
- Wait-list control (No Intervention): Wait-list control of schools without intervention.

INTERVENTIONS:
Behavioral: World Health Organization Health Promoting Schools — Healthy eating: regulation and monitoring of food sold in school cafeterias, healthy eating behavior change campaign, provision of healthy breakfasts.
  Physical activity: hourly active breaks during classes, quality physical education, active recess, and extra-curricular leisure activities and tournaments.
  Healthy hydration: access to water fountains and regular monitoring of water safety, regulation and monitoring of beverages sold in the school, and social marketing campaign promoting drinking plain water.
  Other cross-sectional activities: Referral of children identified as living with underweight, overweight, or obesity, training for school directors, teachers and parents, establishment of school objectives to become a health promoting school, monitoring progress, and publicly acknowledging school progress in becoming a health promoting school.
  Other Names: Salud Escolar; Whole-of-school approach to healthy lifestyles
  Arms: Lifestyle and environment intervention

SUMMARY:
The purpose of this study is to comprehensively evaluate Salud Escolar (School Health), a program led by the Mexican Ministries of Health and Education. This comprehensive evaluation considers a design, implementation, results, and impact evaluation of Salud Escolar.

DETAILED DESCRIPTION:
This study aims is to comprehensively analyze the design, implementation, results, and impact of Salud Escolar, a program led by the Mexican Ministries of Health and Education, during the first phase of implementation, from August 2020 to July 2021. Salud Escolar considers the World Health Organization (WHO) health promoting framework to foster a healthy environment and enhance children's physical activity, healthy eating and hydration. Salud Escolar consists on several activities aligned in the following components: healthy eating, healthy hydration, physical activity and additional cross sectional strategies.

The first phase of implementation will be conducted in a total of 58 schools located in Mexico City purposively selected by the Ministry of Education.

The design evaluation will use available policy documents and program implementation guidelines, scientific literature, to investigate wether the design of Salud Escolar is adequate to achieve the proposed objectives.

The implementation evaluation will be conducted in a sub-sample of 6 intervention schools using qualitative methodologies among key informants.

The results evaluation will be conducted in the 58 intervention schools and pre-post changes in self-reported knowledge, attitudes and practices related to healthy eating, hydration and being physically active will be measured.

The impact evaluation aims to evaluate the effect of Salud Escolar on the consumption of fruits, vegetables and plain water and daily moderate to vigorous physical activity. A sample of 1200 children (6-12 years old) in 15 intervention schools- randomly selected from the sample of 58 intervention schools-, and 15 comparison schools - randomly selected from the waiting list of available schools in the city will be recruited.

Based on the results derived from this analysis, a set of recommendations will be provided to improve the feasibility of scaling up the program at the national level during the second and third phases of Salud Escolar.

ELIGIBILITY:
School

Inclusion criteria:

* Public school
* Minimum of 200 children

Exclusion criteria:

+ None

Children

Inclusion Criteria:

* Aged 6 to 12 years
* Grades 1-6
* Attending school on the day of recruitment at the included schools in Mexico City, Mexico during the school-year 2020/2021

Exclusion Criteria:

+ Schoolchildren with a physical or mental disability not able to participate in daily physical activity or other intervention components or measures.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Physical activity | Change from baseline to 10 months
  Accelerometer-based moderate to vigorous intensity physical activity
Water consumption | Change from baseline to 10 months
  School children's water consumption measured using a 24h dietary recall
Vegetable intake | Change from baseline to 10 months
  School children's vegetable intake measured using a 24h dietary recall
Fruit intake | Change from baseline to 10 months
  School children's fruit intake measured using a 24h dietary recall

SECONDARY OUTCOMES:
Self-reported knowledge | Change from baseline to 10 months
  A questionnaire based on the theory of planned behavior was used to collect relevant knowledge related to healthy eating, drinking plain water and being physically. There are a total of 8 statements and each statement is rated on a 4 point Likert scale. A knowledge score is calculated by estimating the mean score of the responses. Assessed at baseline and 10 months later to estimate change.
Self-reported attitudes | Change from baseline to 10 months
  A questionnaire based on the theory of planned behavior was used to collect relevant attitudes related to healthy eating, drinking plain water and being physically. There are a total of 11 statements and each statement is rated on a 4 point Likert scale. An attitude score is calculated by estimating the mean score of the responses. Assessed at baseline and 10 months later to estimate change.
Perceived behavioral control | Change from baseline to 10 months
  A questionnaire based on the theory of planned behavior is used to collect perceived behavioral control (i.e., self-efficacy) related to healthy eating, drinking plain water and being physically. There are a total of 9 statements and each statement is rated on a 4 point Likert scale. A perceived behavioral control score is calculated by estimating the mean score of the responses. Assessed at baseline and 10 months later to estimate change.
Self-reported physical activity | Change from baseline to 10 months
  The physical activity question of the Health Behaviour in School-aged Children questionnaire is used to rate the proportion of children engaging in at least 60 minutes of moderate to vigorous physical activity per day. Assessed at baseline and 10 months later to estimate change.
Self-reported fruit and vegetable intake | Change from baseline to 10 months
  A questionnaire based on the theory of planned behavior is used to collect practices related to fruit and vegetable intake. There are a total of 3 statements and each statement is rated on a 4 point Likert scale. A fruit and vegetable intake score is calculated by estimating the mean score of the responses. Assessed at baseline and 10 months later to estimate change.
Self-reported junk food intake | Change from baseline to 10 months
  A questionnaire based on the theory of planned behavior is used to collect practices related to junk food consumption (i.e., sweets, candies, pastries, and sugar sweetened beverages). There are a total of 3 statements and each statement is rated on a 4 point Likert scale. A junk food intake score is calculated by estimating the mean score of the responses. Assessed at baseline and 10 months later to estimate change.
Self-reported water consumption | Change from baseline to 10 months
  A questionnaire based on the theory of planned behavior is used to collect practices related to water consumption. There are a total of 2 statements and each statement is rated on a 4 point Likert scale. A water intake score is calculated by estimating the mean score of the responses. Assessed at baseline and 10 months later to estimate change.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Jáuregui, ScD, Principal Investigator — National Institute of public Health
Locations (1):
- Instituto Nacional de Salud Pública, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Data access requests will be reviewed by the principal investigator. Requestors will be required to sign a Data Access agreement.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT04507100/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT04507100/ICF_001.pdf